CLINICAL TRIAL: NCT02998502
Title: Efficacy of a Biofeedback Breathing System for Anxiety and Panic Disorders
Brief Title: The Use of a FDA Cleared, Drug-free, Breathing System for Anxiety and Panic Disorders in Children and Teens
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Palo Alto Health Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB00097094
Record Dates: First submitted 2016-12-09; First posted 2016-12-20 (Estimated); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Anxiety; Panic Disorder
Keywords: Obsessive Compulsive Disorder (OCD); Anxiety; Pediatrics
MeSH Terms: conditions — Anxiety Disorders; Panic Disorder; Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Device Group (Experimental): The Freespira Breathing System (FBS) developed by Palo Alto Health Sciences, Inc, is a portable home device used for breathing biofeedback in adults with PD. FBS has now received FDA clearance for the treatment of PD adults and is currently commercially available and more than 150 therapist have provided the service nationally. However, FBS has not yet been tested for efficacy in a pediatric populations. Due to its portability, FBS may pose an advantage for use in younger age groups, compared to multiple therapy sessions required for CBT or lower acceptability for long-term medication use for adolescent PD. In this pilot intervention study, the efficacy of the FBS system in youth will be tested.
  Interventions: Device: Freespira Breathing System
- Control Group (No Intervention): The device will be given to those in the control group after 8-week baseline period.

INTERVENTIONS:
Device: Freespira Breathing System — Over an 8-week period the efficacy of the FBS system in youth will be tested, with those in the randomized active device group. The control group will not receive the device until completion of the 8 week baseline.
  Arms: Device Group

SUMMARY:
This study will test the efficiency of the Freespira Breathing System in youth.

DETAILED DESCRIPTION:
The Freespira Breathing System (FBS; www.freespira.com) developed by Palo Alto Health Sciences, Inc, is a portable home device , and has been employed in breathing biofeedback in adults with panic disorder (PD). The FBS has now received FDA clearance for the treatment of PD adults and is currently commercially available and more than 150 therapist have provided the service nationally. However, FBS has not yet been tested for efficacy in a pediatric populations. Due to its portability, FBS may pose an advantage for use in younger age groups, compared to multiple therapy sessions required for cognitive behavioral therapy (CBT) or lower acceptability for long-term medication use for adolescent PD.

In this pilot intervention study, the efficacy of the FBS system in youth will be tested. In children adolescents, PD itself is less common than in adults, but when present, PD is commonly associated with and/or preceded by other anxiety conditions, including generalized anxiety disorder (GAD), social phobia (SoP) and separation anxiety (SAD). Thus, in children and adolescents, the breathing biofeedback intervention for panic, should include other anxiety disorders.

ELIGIBILITY:
Inclusion Criteria:

* SCARED score ≥ 25 + prior clinical diagnosis of an anxiety disorder
* Participants must be 9-17 years of age
* If on psychotropic medication(s), participant must be on a stable dose for at least one month prior to study enrollment

Exclusion Criteria:

* Anxiety has occurred exclusively during a major depressive episode, psychiatric illness, dementia, intellectual disability, or brain disease
* Currently enrolled in another device or drug study or less than 30 days has elapsed since participation in such a study
* Currently undergoing breathing biofeedback elsewhere
* Demonstrate evidence of severe suicidal ideation or psychosis
* There is an active condition of asthma

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 73 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Screen for Child Anxiety Related Disorders (SCARED) scale score | 8-weeks
  The Screen for Child Anxiety Related Disorders (SCARED) is a 41-item inventory rated on a 3 point Likert-type scale. It comes in two versions; one asks questions to parents about their child and the other asks these same questions to the child directly. The purpose of the instrument is to screen for signs of anxiety disorders in children.

SECONDARY OUTCOMES:
SCARED anxiety scale score | Baseline
  The Screen for Child Anxiety Related Disorders (SCARED) is a 41-item inventory rated on a 3 point Likert-type scale. It comes in two versions; one asks questions to parents about their child and the other asks these same questions to the child directly. The purpose of the instrument is to screen for signs of anxiety disorders in children.
SCARED anxiety scale score | Week 4 Follow Up
  The Screen for Child Anxiety Related Disorders (SCARED) is a 41-item inventory rated on a 3 point Likert-type scale. It comes in two versions; one asks questions to parents about their child and the other asks these same questions to the child directly. The purpose of the instrument is to screen for signs of anxiety disorders in children.
SCARED anxiety scale score | Week 8 Follow Up
  The Screen for Child Anxiety Related Disorders (SCARED) is a 41-item inventory rated on a 3 point Likert-type scale. It comes in two versions; one asks questions to parents about their child and the other asks these same questions to the child directly. The purpose of the instrument is to screen for signs of anxiety disorders in children.
SCARED anxiety scale score | 6-month Follow Up
  The Screen for Child Anxiety Related Disorders (SCARED) is a 41-item inventory rated on a 3 point Likert-type scale. It comes in two versions; one asks questions to parents about their child and the other asks these same questions to the child directly. The purpose of the instrument is to screen for signs of anxiety disorders in children.
SCARED anxiety scale score | 12-month Follow Up
  The Screen for Child Anxiety Related Disorders (SCARED) is a 41-item inventory rated on a 3 point Likert-type scale. It comes in two versions; one asks questions to parents about their child and the other asks these same questions to the child directly. The purpose of the instrument is to screen for signs of anxiety disorders in children.
End-tidal carbon dioxide (CO2) | 4 weeks
  End-tidal CO2 at 4 weeks Measured using Freespira breathing system 4 minutes breathing session Parameters number of millimeters per mercury.
Respiratory rate level | 4 weeks
  Respiratory rate at 4 weeks Measured using Freespira breathing system 4 minutes breathing session. The parameters are number of breaths per minute.
Panic Disorder Severity Scale for Adolescents (PDSS-A) | Baseline
  Panic Disorder Severity Scale for Adolescents [PDSS-A] seven question scale referring to panic attacks and symptoms during each episode and how severe the attacks were. Each question is given a rating from 0-4 and the total score from each of the seven questions becomes the score used to assess severity. The higher the score the more severe the panic disorder.
Panic Disorder Severity Scale for Adolescents (PDSS-A) | Week 4 Follow Up
  Panic Disorder Severity Scale for Adolescents [PDSS-A] seven question scale referring to panic attacks and symptoms during each episode and how severe the attacks were. Each question is given a rating from 0-4 and the total score from each of the seven questions becomes the score used to assess severity. The higher the score the more severe the panic disorder.
Panic Disorder Severity Scale for Adolescents (PDSS-A) | Week 8 Follow Up
  Panic Disorder Severity Scale for Adolescents [PDSS-A] seven question scale referring to panic attacks and symptoms during each episode and how severe the attacks were. Each question is given a rating from 0-4 and the total score from each of the seven questions becomes the score used to assess severity. The higher the score the more severe the panic disorder.
Panic Disorder Severity Scale for Adolescents (PDSS-A) | 6-Month Follow Up
  Panic Disorder Severity Scale for Adolescents [PDSS-A] seven question scale referring to panic attacks and symptoms during each episode and how severe the attacks were. Each question is given a rating from 0-4 and the total score from each of the seven questions becomes the score used to assess severity. The higher the score the more severe the panic disorder.
Panic Disorder Severity Scale for Adolescents (PDSS-A) | 12 month Follow Up
  Panic Disorder Severity Scale for Adolescents [PDSS-A] seven question scale referring to panic attacks and symptoms during each episode and how severe the attacks were. Each question is given a rating from 0-4 and the total score from each of the seven questions becomes the score used to assess severity. The higher the score the more severe the panic disorder.
Clinician's Global Impression scale. | Baseline
  Clinician's Global Impression (CGI) scale is a three item observer rated scale that measures illness severity, global improvement or change, and therapeutic response. It is rated on a seven point scale with the severity of illness scale using a range of responses from one (normal) to seven (around the most severely ill patients). Each component of the CGI is rated separately; the instrument does not yield a global score.
  This will serve as the measure of overall improvement in the patients symptoms because of the FBS treatment.
Clinician's Global Impression scale. | Week 4 Follow Up
  Clinician's Global Impression (CGI) scale is a three item observer rated scale that measures illness severity, global improvement or change, and therapeutic response. It is rated on a seven point scale with the severity of illness scale using a range of responses from one (normal) to seven (around the most severely ill patients). Each component of the CGI is rated separately; the instrument does not yield a global score.
  This will serve as the measure of overall improvement in the patients symptoms because of the FBS treatment.
Clinician's Global Impression scale. | Week 8 Follow Up
  Clinician's Global Impression (CGI) scale is a three item observer rated scale that measures illness severity, global improvement or change, and therapeutic response. It is rated on a seven point scale with the severity of illness scale using a range of responses from one (normal) to seven (around the most severely ill patients). Each component of the CGI is rated separately; the instrument does not yield a global score.
  This will serve as the measure of overall improvement in the patients symptoms because of the FBS treatment.
Child Yale Brown Obsessive-Compulsive Scale score | Baseline
  Child Yale Brown Obsessive-Compulsive Scale is a measure of obsessive compulsion disorder symptoms. This scale is designed to rate the severity of obsessive and compulsive symptoms in children from 6-17 years. In general the ratings depend on the child's and parents report; however the final rating is based on the clinical judgement of the interviewer. The characteristics of each item over the prior week up until; and including, the time of the interview are rated. The child's symptoms are scored using the compulsions checklist and the obsessions checklist as guides. All 19 items are rated but only items 1-10 are used to determine the final score. The total score is the sum of items 1-10; the obsession and compulsion subtotals are the sums of items 1-5 and 6-10, respectively. This will be measured through out the study to see the effectiveness of the treatment.
Child Yale Brown Obsessive-Compulsive Scale score | Week 4 Follow Up
  Child Yale Brown Obsessive-Compulsive Scale is a measure of obsessive compulsion disorder symptoms. This scale is designed to rate the severity of obsessive and compulsive symptoms in children from 6-17 years. In general the ratings depend on the child's and parents report; however the final rating is based on the clinical judgement of the interviewer. The characteristics of each item over the prior week up until; and including, the time of the interview are rated. The child's symptoms are scored using the compulsions checklist and the obsessions checklist as guides. All 19 items are rated but only items 1-10 are used to determine the final score. The total score is the sum of items 1-10; the obsession and compulsion subtotals are the sums of items 1-5 and 6-10, respectively. This will be measured through out the study to see the effectiveness of the treatment.
Child Yale Brown Obsessive-Compulsive Scale score | Week 8 Follow Up
  Child Yale Brown Obsessive-Compulsive Scale is a measure of obsessive compulsion disorder symptoms. This scale is designed to rate the severity of obsessive and compulsive symptoms in children from 6-17 years. In general the ratings depend on the child's and parents report; however the final rating is based on the clinical judgement of the interviewer. The characteristics of each item over the prior week up until; and including, the time of the interview are rated. The child's symptoms are scored using the compulsions checklist and the obsessions checklist as guides. All 19 items are rated but only items 1-10 are used to determine the final score. The total score is the sum of items 1-10; the obsession and compulsion subtotals are the sums of items 1-5 and 6-10, respectively. This will be measured through out the study to see the effectiveness of the treatment.
Decrease in severity of panic attacks as documented in panic dairy (only for participants with panic attacks) | Week 8
  Decrease in severity of panic attacks as documented in panic dairy (only for participants with panic attacks)

OTHER OUTCOMES:
Child Sheehan Disability Scale (CSDS) | Baseline
  The CSDS was designed to measure the extent to which the child's anxiety symptoms were interfering with daily functioning. The CSDS is an adaptation of the Sheehan Disability Scale and consisted of items inquiring about the degree to which the child's anxiety symptoms interfere with school, social, and family functioning. As on the SDS, items are measured on an 11-point Likert-type scale ranging from 0 (not at all) to 10 (very, very much) .The wording of the anchors on the SDS was adapted to be more appropriate for children. A parent version (CSDS-P) that included six items was also created. The CSDS-P included three items that assessed the degree to which the parents perceived the child's anxiety symptoms to be interfering with the child's functioning (school, social, family) as well as three items that assessed the degree to which the child's symptoms were viewed as interfering with the parent's functioning (work, social, family).
Child Sheehan Disability Scale (CSDS) | Week 4 Follow Up
  The CSDS was designed to measure the extent to which the child's anxiety symptoms were interfering with daily functioning. The CSDS is an adaptation of the Sheehan Disability Scale and consisted of items inquiring about the degree to which the child's anxiety symptoms interfere with school, social, and family functioning. As on the SDS, items are measured on an 11-point Likert-type scale ranging from 0 (not at all) to 10 (very, very much) .The wording of the anchors on the SDS was adapted to be more appropriate for children. A parent version (CSDS-P) that included six items was also created. The CSDS-P included three items that assessed the degree to which the parents perceived the child's anxiety symptoms to be interfering with the child's functioning (school, social, family) as well as three items that assessed the degree to which the child's symptoms were viewed as interfering with the parent's functioning (work, social, family).
Child Sheehan Disability Scale (CSDS) | Week 8 Follow Up
  The CSDS was designed to measure the extent to which the child's anxiety symptoms were interfering with daily functioning. The CSDS is an adaptation of the Sheehan Disability Scale and consisted of items inquiring about the degree to which the child's anxiety symptoms interfere with school, social, and family functioning. As on the SDS, items are measured on an 11-point Likert-type scale ranging from 0 (not at all) to 10 (very, very much) .The wording of the anchors on the SDS was adapted to be more appropriate for children. A parent version (CSDS-P) that included six items was also created. The CSDS-P included three items that assessed the degree to which the parents perceived the child's anxiety symptoms to be interfering with the child's functioning (school, social, family) as well as three items that assessed the degree to which the child's symptoms were viewed as interfering with the parent's functioning (work, social, family).
Children's Depression Inventory ( CDI2) | Baseline
  The Children's Depression Inventory (CDI and CDI2) is a psychological assessment that rates the severity of symptoms related to depression or dysthymic disorder in children and adolescents. The CDI is a 27-item scale that is self-rated and symptom-oriented. The assessment is now in its second edition. The 27 items on the assessment are grouped into five major factor areas. Clients rate themselves based on how they feel and think, with each statement being identified with a rating from 0 to 2.
Children's Depression Inventory ( CDI2) | Week 4 Follow Up
  The Children's Depression Inventory (CDI and CDI2) is a psychological assessment that rates the severity of symptoms related to depression or dysthymic disorder in children and adolescents. The CDI is a 27-item scale that is self-rated and symptom-oriented. The assessment is now in its second edition. The 27 items on the assessment are grouped into five major factor areas. Clients rate themselves based on how they feel and think, with each statement being identified with a rating from 0 to 2.
Children's Depression Inventory ( CDI2) | Week 8 Follow Up
  The Children's Depression Inventory (CDI and CDI2) is a psychological assessment that rates the severity of symptoms related to depression or dysthymic disorder in children and adolescents. The CDI is a 27-item scale that is self-rated and symptom-oriented. The assessment is now in its second edition. The 27 items on the assessment are grouped into five major factor areas. Clients rate themselves based on how they feel and think, with each statement being identified with a rating from 0 to 2.
Childhood Anxiety Sensitivity Index (CASI) | Baseline
  The Child Anxiety Sensitivity Index is an 18-item scale which measures anxiety sensitivity by asking children to state how aversely they view anxiety symptoms. The child is to mark either "none" (I), "some" (2), or "A Lot" (3) to each item. The child's total anxiety sensitivity score is the sum of his or her points.
Childhood Anxiety Sensitivity Index (CASI) | Week 4 Follow Up
  The Child Anxiety Sensitivity Index is an 18-item scale which measures anxiety sensitivity by asking children to state how aversely they view anxiety symptoms. The child is to mark either "none" (I), "some" (2), or "A Lot" (3) to each item. The child's total anxiety sensitivity score is the sum of his or her points.
Childhood Anxiety Sensitivity Index (CASI) | Week 8 Follow Up
  The Child Anxiety Sensitivity Index is an 18-item scale which measures anxiety sensitivity by asking children to state how aversely they view anxiety symptoms. The child is to mark either "none" (I), "some" (2), or "A Lot" (3) to each item. The child's total anxiety sensitivity score is the sum of his or her points.
Junior Temperament and Character Inventory (JTCI) | Baseline
  The Junior Temperament and Character Inventory (JTCI) was developed to assess the temperament ('novelty seeking', 'harm avoidance', 'reward dependence', 'persistence') and character ('self-directedness', 'cooperativeness', 'self-transcendence') dimensions of Cloninger's bio-social model of personality in children and adolescents. Each of the 108 statements can be answered "True" or "False". The parent is to decide which choice best fits the child they are describing in this questionnaire.
Kiddie Schedule for Affective Disorders and Schizophrenia (K-SADS) | Baseline
  The Kiddie Schedule for Affective Disorders and Schizophrenia (K-SADS) is a semi-structured interview aimed at early diagnosis of affective disorders such as depression, bipolar disorder, and anxiety disorder. There are currently four different versions of the test that are structured to include interviews with both the child and the parents or guardians.
Kiddie Schedule for Affective Disorders and Schizophrenia (K-SADS) | Week 4 Follow Up
  The Kiddie Schedule for Affective Disorders and Schizophrenia (K-SADS) is a semi-structured interview aimed at early diagnosis of affective disorders such as depression, bipolar disorder, and anxiety disorder. There are currently four different versions of the test that are structured to include interviews with both the child and the parents or guardians.
Kiddie Schedule for Affective Disorders and Schizophrenia (K-SADS) | Week 8 Follow Up
  The Kiddie Schedule for Affective Disorders and Schizophrenia (K-SADS) is a semi-structured interview aimed at early diagnosis of affective disorders such as depression, bipolar disorder, and anxiety disorder. There are currently four different versions of the test that are structured to include interviews with both the child and the parents or guardians.
Kiddie Schedule for Affective Disorders and Schizophrenia (K-SADS) | 12 month Follow Up
  The Kiddie Schedule for Affective Disorders and Schizophrenia (K-SADS) is a semi-structured interview aimed at early diagnosis of affective disorders such as depression, bipolar disorder, and anxiety disorder. There are currently four different versions of the test that are structured to include interviews with both the child and the parents or guardians.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Grados, M.D., M.P.H., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-17): https://cdn.clinicaltrials.gov/large-docs/02/NCT02998502/Prot_SAP_001.pdf
  • Informed Consent Form (2017-11-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT02998502/ICF_000.pdf